CLINICAL TRIAL: NCT03368768
Title: Antibiotic Footprint Thailand - Pilot Questionnaire Study
Acronym: AFT PILOT
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO1704
Record Dates: First submitted 2017-10-30; First posted 2017-12-11 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Antibiotic Usage
Keywords: Antimicrobial-resistant bacterial infection; Questionaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Contact group email of Mahidol-Oxford Research Unit (MORU): The investigator aims to have at least 100 adult people who could provide information for the total of one year. This expects that at least 20 of those 100 people would have common cold or diarrhea at least one time over one year period. This should provide more than 80% power to detect whether the proportion of having antibiotics when they have common cold or diarrhea was lower than 50% or not. The hypothesized proportion was 20% as stated by the national strategy against AMR in Thailand
  Interventions: Other: Obtain inform consent via questionnaire of Monkey Survey

INTERVENTIONS:
Other: Obtain inform consent via questionnaire of Monkey Survey — This is an internet-based questionnaire study. Therefore, anyone in Thailand can access and answer the questionnaire.

SUMMARY:
Antimicrobial-resistant bacterial infection is an important cause of death in Thailand and in other countries worldwide. Increasing use of antibiotics in both animals and humans is one of the main drive that increase the incidence of antimicrobial resistant bacteria in human, animals and environment.

National Action Plan for Combating Antibiotic-resistant Bacteria aimed to have general population taking antibiotics less than 20% when they have common cold or diarrheal symptoms. However, there is little accurate information about behaviors of Thai people. Most studies were conducted in hospitals, clinics or pharmacy. Therefore, it did not include behaviors of those who had symptoms but did not present at hospitals, clinics or pharmacy.

In this study, the investigators aim to use questionnaire to Thai adult population to ask for the the amount of antibiotic used and the periods they had symptoms of common cold or diarrhea over one year period of year 2017. The main aim is to estimate the total antibiotic usage per human population, and plan for the study in the future.

ELIGIBILITY:
Inclusion Criteria:

The participant may enter the study if ALL of the following apply:

1. Participant is willing and able to give informed consent for participation in the study.
2. Male or female, aged 18 years or above.
3. Living in Thailand (staying in Thailand more than 6 months per year)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Living in Thailand (staying in Thailand more than 6 months per year)
Study Population: This study aims to have at least 100 adult people who could provide information for the total of one year. This expects that at least 20 of those 100 people would have common cold or diarrhea at least one time over one year period. This should provide more than 80% power to detect whether the proportion of having antibiotics when they have common cold or diarrhea was lower than 50% or not. The hypothesizjed proportion was 20% as stated by the national strategy against AMR in Thailand.
  MORU has a total number of staff for more than 200 people, and we suspect that the internal people in MORU should be enough for the study. We will also want to pilot whether the internet-based study can spread into the community well or not.
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Total antibiotic usage in human population | 1 year

SECONDARY OUTCOMES:
Association between the antibiotic usage and the episodes of common cold | 1 year
  Association between the antibiotic usage and the episodes of common cold or diarrhea in Thai adult population
Association between the antibiotic usage and the episodes of diarrhea | 1 year
  Association between the antibiotic usage and the episodes of common cold or diarrhea in Thai adult population

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol-Oxford Tropical Medicine Research Unit (MORU), Faculty of Tropical Medicine, Mahidol University, Thailand, Bangkok, Thailand